CLINICAL TRIAL: NCT06661629
Title: Characterizing Bilateral Hypoglossal Nerve Stimulation During Drug-Induced Sleep Endoscopy (BLISS - BiLateral Inspire Sedated Stimulation)
Brief Title: Characterizing Bilateral Hypoglossal Nerve Stimulation During Drug-Induced Sleep Endoscopy
Acronym: BLISS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prior to enrollment following mutual agreement between the sponsor and the site. No patients were recruited. No data was collected.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25477
Record Dates: First submitted 2024-10-16; First posted 2024-10-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: OSA - Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral vs Bilateral HGNS (Experimental): All participants will undergo both unilateral and bilateral hypoglossal nerve stimulation during a single drug-induced sleep endoscopy exam. The voltage will be adjusted [0.1 5.0 V].
  Interventions: Device: Nerve stimulation

INTERVENTIONS:
Device: Nerve stimulation — The intervention is testing the effect of unilateral versus bilateral hypoglossal nerve stimulation on upper airway collapsibility during drug-induced sleep endoscopy

SUMMARY:
The study will investigate the treatment effect of bilateral genioglossus muscle stimulation on upper airway collapsibility during drug-induced sleep endoscopy in patients implanted with the Inspire hypoglossal nerve stimulator.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 22yrs) willing and capable of providing informed consent
* Implanted with the Inspire hypoglossal nerve stimulator

Exclusion Criteria:

* • Pregnant women*

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Upper Airway Collapsability Measures | During DISE - during the 20 minutes that the Drug Induced Sleep Endoscopy Occurs.
  PhOP - Pharangeal Opening Pressure, the minimum CPAP level needed to have an unobstructed airway
Upper Airway Collapsability Measures | During DISE - during the 20 minutes that the Drug Induced Sleep Endoscopy Occurs
  Pcrit - Critical Pressure, the maximum CPAP level where the airway is obstructed

SECONDARY OUTCOMES:
Difference in Voltage Requirements | During DISE - During the 20 minutes during which the Drug Induced Sleep Endoscopy occurs
  Difference in voltage between Inspire Device and External Stimulator during unilateral and bilateral stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Raj C Dedhia, MD, Principal Investigator — Penn Medicine

IPD SHARING:
Plan to Share IPD: Yes
CTA is being drafted for data sharing between Penn Medicine and Inspire Medical Systems - IPD would be shared between Penn and Inspire.
Supporting Information: Study Protocol, SAP, ICF